CLINICAL TRIAL: NCT05995327
Title: Construction of an Ambispective Cohort for Unplanned Spinal Re-operation
Brief Title: Reasons and Risk Factors for Unplanned Spinal Re-operation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: PUTH Beifang Hospital (Unknown); PUTH Chongli Hospital (Unknown); PUTH Qinhuangdao Hospital (Unknown); PUTH Yanqing Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: M2022045
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Degeneration Spine; Spine Deformity; Spine Tumor; Spine Fracture
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- spine degenerative disease: patients with spine degenerative disease
- spine tumor: patients with spinal tumors
- spine deformity: patients with spinal deformity
- spine fracture: patients with spine fracture

SUMMARY:
Unplanned re-operation is one of the common negative indicators reflecting the quality and safety of surgery in the medical industry and has become one of the ten goals for the improvement of national medical quality and safety in China since 2022, while about 40% of unplanned re-operations in Peking University Third Hospital in recent years occur in spine patients of the orthopedics department. This project intends to establish a high-quality and sustainable ambispective disease cohort for spine surgery in Peking University Third Hospital based on the unplanned re-operations that occurred in the Orthopedics Department of Peking University Third Hospital from January 2012 to December 2025. The investigators further summarize and analyze clinical causes and risk factors of re-operations, aiming to explore scientific coping strategies and provide reference for continuous improvement of medical service quality.

DETAILED DESCRIPTION:
Unplanned re-operation is one of the common negative indicators reflecting the quality and safety of surgery in the medical industry. Possible reasons for a patient's return to the operating room include problems with surgical technique, anesthesia procedures, or infection control. Reducing the rate of unplanned re-operation has become one of the ten goals for the improvement of national medical quality and safety in China since 2022, and has been paid more and more attention by the National Health Commission and hospital managers.

About 40% of the unplanned re-operations in Peking University Third Hospital in recent years occur in spine patients of the orthopedics department, thus lowering the rate of spine unplanned re-operations is of great significance to improve the overall medical quality and safety. Driven by the common needs and joint force of "nation-hospital-department", this project intends to establish a high-quality and sustainable ambispective disease cohort for spine surgery in Peking University Third Hospital based on unplanned re-operations that occurred in the Orthopedics Department of Peking University Third Hospital from January 2012 to December 2025. The investigators further summarize and analyze clinical causes and risk factors of re-operations, aiming to explore scientific coping strategies and provide reference for continuous improvement of medical service quality. Furthermore, the investigators intend to construct multiple risk prediction models for spine unplanned re-operation and special disease cohorts. This project will form a synergy in the three aspects of "clinical, scientific research, and management", lower the unplanned re-operation rate of orthopedic spinal surgery, improve medical quality and safety management in Peking University Third Hospital, and promote the in-depth exploration and vigorous development of spine discipline in the scientific fields of perioperative safety and risk assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received orthopedic surgery in Peking University Third Hospital, including spinal degeneration, spinal deformity, spinal tumor, spine fracture reduction and internal fixation
2. Both the initial surgery and unplanned re-operation were completed in the orthopedic department of Peking University Third Hospital
3. The interval between two surgeries is within 30 days
4. Discharged from the orthopedics department of Peking University Third Hospital

Exclusion Criteria:

1. Re-operation for other systemic diseases unrelated to the initial surgery
2. Re-operation is a clinical procedure that is not a return to the operating room, such as wound debridement and suturing, skull traction, etc. performed in the ward

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the retrospective cohort, patients were enrolled from January 2012 to December 2021. They aged from 18 to 80 years with spinal disease who were hospitalized for surgery in the orthopedics department of Peking University Third Hospital and had complete medical records, while diagnosing of fracture, limb arthritis, limb tumor and other non-spinal diseases were excluded.
  In the prospective cohort, patients were enrolled from January 2023 to December 2025; They aged from 18 to 80 years with spinal disease who were hospitalized for surgery in the orthopedics department of Peking University Third Hospital, while diagnosing of fracture, limb arthritis, limb tumor and other non-spinal diseases were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 70000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of spine unplanned re-operation | 30 days
  We calculate the unplanned re-operation incidences in total and that of specialized spinal diseases.

SECONDARY OUTCOMES:
reasons of spine unplanned re-operation | 30 days
  We summarize reasons of spine unplanned re-operation in total and that of specialized spinal diseases.
risk factors of spine unplanned re-operation | 30 days
  We figure out risk factors of spine unplanned re-operation and that of specialized spinal diseases by comparing conditions between patients underwent unplanned re-operation or not.

CONTACTS AND LOCATIONS:
Overall Officials: Weishi Li, Study Chair — Peking University Third Hospital
Locations (5):
- China (5):
  - PUTH Beifang Hospital, Beijing
  - PUTH Chongli Hospital, Beijing
  - PUTH Qinhuangdao Hospital, Beijing
  - PUTH Yanqing Hospital, Beijing
  - Peking University Third Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ouyang H, Hu Y, Hu W, Zhang H, Sun Z, Tang Y, Jiang Y, Chen J, Dong S, Li W, Tian Y. Incidences, causes and risk factors of unplanned reoperations within 30 days of spine surgery: a single-center study based on 35,246 patients. Spine J. 2022 Nov;22(11):1811-1819. doi: 10.1016/j.spinee.2022.07.098. Epub 2022 Jul 22. PMID 35878756
- [Result] Hu Y, Ouyang H, Ye K, Qi J, Dong Y, Peng X, Zhang X, Dong S, Chen Z, Liu Z, Liu X, Sun C, Li W, Tian Y. Thirty-day Unplanned Reoperations After Posterior Surgery for Thoracic Spinal Stenosis: A Single-center Study Based on 1948 Patients. Spine (Phila Pa 1976). 2023 Apr 1;48(7):507-513. doi: 10.1097/BRS.0000000000004499. Epub 2022 Oct 3. PMID 36191058
- [Result] Hu Y, Ouyang H, Ye K, Dong Y, Zhang X, Dong S, Chen Z, Liu Z, Liu X, Zeng Y, Wei F, Sun C, Tian Y, Li W. Thirty-day unplanned reoperations of thoracic spine surgery: 10 years of data from a single center with 3242 patients. Spine J. 2023 May;23(5):703-714. doi: 10.1016/j.spinee.2023.01.005. Epub 2023 Jan 11. PMID 36641036